CLINICAL TRIAL: NCT06991959
Title: Can Education for Rural Women Lift the Fog Behind Closed Doors?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Burcu KUCUKKAYA, Asst. Prof, Bartın Unıversity
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2024-SBB-0313
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Contraception; Sexually Transmitted Diseases
Keywords: Rural; Education; Knowledge; Attitudes
MeSH Terms: conditions — Sexually Transmitted Diseases; Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Education (Experimental)
  Interventions: Other: Educaton

INTERVENTIONS:
Other: Educaton — Family Planning and Sexually Transmitted Diseases Training: The training program used a training module developed by UNFPA based on health belief theory, theory of reason-based behavior, social learning theory and transtheoretical model.
  Arms: Education

SUMMARY:
The aim of this study was to investigate the effect of family planning and sexually transmitted diseases education given to rural women on their level of knowledge and attitudes towards reproductive health and family planning. Design: The prospective, randomized controlled study

ELIGIBILITY:
Inclusion Criteria:

* Women who can speak Turkish,
* Are older than 18 years of age,
* Do not have a diagnosis of hearing impairment,
* Live with their husband/partner,
* Have an active sexual life,
* Live in the districts within the borders of Bartın province,
* Do not have a type of cancer that may affect sexual function,
* Have not received family planning and sexually transmitted diseases training before,
* Have written informed consent,
* Volunteer to participate in the study

Exclusion Criteria:

* Women who received family planning and sexually transmitted diseases education from another counselor during the study period,
* Did not participate in the post-test,
* Did not volunteer to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 72 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Sexually Transmitted Diseases Knowledge Scale | change from before implamentation patent and after 1st day of practice.
  The 25-item, 6-sub-dimensional STIPS was found to be acceptably compatible with Turkish culture. Correct answers to each item in the scale are worth 1 point, while incorrect or don't know answers are worth 0 points. The highest total score to be obtained from the scale is 25 and the lowest score is 0.
Reproductive Health and Family Planning Attitude Scale | change from before implamentation patent and after 1st day of practice.
  The scale has 3 sub-dimensions: 'unwanted pregnancies', 'sexually transmitted infections' and 'infertility and fertility treatments'. The scale has no cut-off point. As the score obtained from the scale increases, attitudes towards reproductive health and FP become more positive. The highest score that can be obtained from the scale is 5. Cronbach's alpha of the scale is 0.88.

CONTACTS AND LOCATIONS:
Locations (1):
- Bartın University, Bartın, Turkey (Türkiye)